CLINICAL TRIAL: NCT04858412
Title: Evaluate the Molecular Mechanisms of HMB-enriched Amino Acid Supplement to Reverse Muscle Loss in Patients With Alcoholic Liver Disease and COVID-19
Brief Title: Study of HMB-enriched Amino Acid Supplementation in Patients With Alcoholic Liver Disease and COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Srinivasan Dasarathy, Staff, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 20-1194
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Alcoholic Liver Disease; COVID 19 Pneumonia
MeSH Terms: conditions — Liver Diseases, Alcoholic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HMB enriched amino acid arm (Active Comparator): The patients randomized to the HMB enriched amino acid (HMB/EAA) arm will be given HMB/EAA for 90 days.
  Interventions: Dietary Supplement: β-hydroxy β-methyl butyrate (HMB) enriched amino acid
- Balanced amino acid arm (Placebo Comparator): The patients randomized to the Balanced amino acid (BAA) arm will be given BAA for 90 days.
  Interventions: Dietary Supplement: Balanced amino acid

INTERVENTIONS:
Dietary Supplement: β-hydroxy β-methyl butyrate (HMB) enriched amino acid — β-hydroxy β-methyl butyrate (HMB) is a non-nitrogenous leucine metabolite with anabolic properties.
  Arms: HMB enriched amino acid arm
Dietary Supplement: Balanced amino acid — Balanced amino acid is the balanced mixture of the various essential amino acids.
  Arms: Balanced amino acid arm

SUMMARY:
Patients with COVID-19 and comorbidities including alcohol associated liver disease (ALD) are at risk for severe illness and abrupt or sudden clinical deterioration with ventilatory failure. â-hydroxy â-methyl butyrate (HMB), a non-nitrogenous leucine metabolite with anabolic properties, increases muscle mass and contractile function and enhances immune function. We aim to study the natural course of COVID-19 in patients with ALD and test whether HMB can affect ventilatory deterioration and improve short and long-term morbidity, mortality, and recovery from critical illness in symptomatic COVID-19 patients with ALD.

ELIGIBILITY:
Inclusion Criteria:

A. Cases: Patients with ALD and COVID-19 pneumonia:

1. Clinical, imaging, laboratory, and/or histological diagnosis of alcoholic cirrhosis and/or alcoholic hepatitis
2. Child Pugh score 5-8, serum creatinine <3, Model for End Stage Liver Disease score (MELD) <25
3. Diagnosis of COVID-19 pneumonia as defined by the WHO criteria: confirmed SARS-CoV-2 infection by PCR, evidence of bilateral pulmonary infiltrates on chest radiograph (CXR) or computed tomography (CT) and SpO2 <93% or on oxygen supplement
4. Age of 21 years or older

B. Controls: Patients without alcoholic liver disease (Non-ALD) and COVID-19 pneumonia:

1. Diagnosis of COVID-19 pneumonia as defined by the WHO criteria: confirmed SARS-CoV-2 infection by PCR, evidence of bilateral pulmonary infiltrates on chest radiograph (CXR) or computed tomography (CT) and SpO2 <93% or on oxygen supplement
2. Age of 21 years or older

Exclusion Criteria: (Both Cases and Controls)

1. Patients requiring active ventilator support
2. Anticoagulant/antiplatelet therapy (for those in the biopsy arm, see Randomization schema. If clinically feasible, patients will be asked to hold their anticoagulants for the muscle biopsy after physician review),
3. Recent gastrointestinal bleeding (<3 months)
4. Advanced organ diseases: congestive heart failure (NYHA class 3 and 4), chronic obstructive pulmonary diseases (COPD) (GOLD stage 3 and 4), chronic kidney disease (Cr>3), metastatic malignancy
5. Medications that alter muscle protein metabolism except systemic corticosteroids
6. Pregnancy
7. Unwillingness/ Inability to sign informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in skeletal muscle mass at Day 0 and Day 90 | Baseline and Day 90
Number of hospital admissions between Day 0 and Day 90 | Baseline and Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Dasarathy, MD, Principal Investigator — Staff
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No